CLINICAL TRIAL: NCT00227227
Title: Observational Study With Enbrel (Etanercept) in Patients With Ankylosing Spondylitis
Brief Title: Study Evaluating Enbrel (Etanercept) in Patients With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 101540
Record Dates: First submitted 2005-09-13; First posted 2005-09-27 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate the incidence of adverse events for patients with AS treated with Enbrel in usual care settings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis

Exclusion Criteria:

* Contraindications according SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2004-05; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — MedinfoDEU@wyeth.com
Locations (1):
- Berlin, Germany